CLINICAL TRIAL: NCT07289620
Title: A Randomized, Double-Blinded, Controlled Trial Comparing Perineural Dexamethasone, Dexmedetomidine, and Their Combination as Adjuvants to Ropivacaine for Popliteal Sciatic Nerve Block in Pediatric Patients
Brief Title: Dexamethasone vs Dexmedetomidine vs Combination as Adjuvants to Popliteal Sciatic Nerve Block in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Ankle Disease; Foot Diseases
MeSH Terms: conditions — Foot Diseases | interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perineural Dexamethasone (Active Comparator): Children in this arm will receive a single-shot popliteal sciatic nerve block performed under ultrasound guidance with 0.3 mL/kg of 0.2% ropivacaine combined with 0.1 mg/kg perineural dexamethasone (maximum dose per institutional pediatric guidelines). The block will be performed using a 22-gauge echogenic needle under sterile conditions prior to the start of surgery. No additional adjuvants will be administered. Standard perioperative analgesia will be provided to all participants.
  Interventions: Drug: Dexamethasone
- Perineural Dexmedetomidine (Active Comparator): Children in this arm will receive a single-shot popliteal sciatic nerve block performed under ultrasound guidance with 0.3 mL/kg of 0.2% ropivacaine combined with 0.5 µg/kg perineural dexmedetomidine (maximum dose per institutional pediatric guidelines). A 22-gauge echogenic needle will be used for block placement under sterile conditions. No additional adjuvants will be administered. Standard perioperative analgesia will be provided to all participants.
  Interventions: Drug: Dexmedetomidine
- Perineural Dexamethasone + Dexmedetomidine Combination (Active Comparator): Children in this arm will receive a single-shot popliteal sciatic nerve block performed under ultrasound guidance with 0.3 mL/kg of 0.2% ropivacaine combined with 0.1 mg/kg perineural dexamethasone and 0.5 µg/kg perineural dexmedetomidine (maximum doses per institutional pediatric guidelines). The block will be performed with a 22-gauge echogenic needle under sterile conditions before surgery. Standard perioperative analgesia will be provided to all participants.
  Interventions: Drug: Dexamethasone + Dexmedetomidine

INTERVENTIONS:
Drug: Dexamethasone — Perineural dexamethasone will be administered as an adjuvant to a single-shot popliteal sciatic nerve block. Children will receive 0.3 mL/kg of 0.2% ropivacaine combined with 0.1 mg/kg dexamethasone, injected under ultrasound guidance using a 22-gauge echogenic needle prior to surgery. The medication will be given as a single perineural dose only. Standard perioperative analgesia will be provided to all participants.
  Arms: Perineural Dexamethasone
Drug: Dexmedetomidine — Perineural dexmedetomidine will be administered as an adjuvant to a single-shot popliteal sciatic nerve block. Children will receive 0.3 mL/kg of 0.2% ropivacaine combined with 0.5 µg/kg dexmedetomidine, injected under ultrasound guidance with a 22-gauge echogenic needle prior to surgery. The medication will be administered as a single perineural bolus. Standard perioperative analgesia will be provided to all participants.
  Arms: Perineural Dexmedetomidine
Drug: Dexamethasone + Dexmedetomidine — Children in this arm will receive a combination of two perineural adjuvants added to a single-shot popliteal sciatic nerve block. The block will include 0.3 mL/kg of 0.2% ropivacaine combined with 0.1 mg/kg dexamethasone and 0.5 µg/kg dexmedetomidine, administered under ultrasound guidance using a 22-gauge echogenic needle prior to surgery. Both medications will be delivered together as a single perineural bolus. Standard perioperative analgesia will be provided to all participants.
  Arms: Perineural Dexamethasone + Dexmedetomidine Combination

SUMMARY:
This clinical study will evaluate three commonly used medications that can be added to local anesthetic during a popliteal sciatic nerve block in children undergoing surgery of the lower leg or foot. These medications-dexamethasone, dexmedetomidine, or a combination of both-may help the nerve block last longer and provide better postoperative pain control.

All participating children will receive a standard popliteal sciatic nerve block with ropivacaine, a commonly used local anesthetic. They will then be randomly assigned to one of three groups: (1) ropivacaine with dexamethasone, (2) ropivacaine with dexmedetomidine, or (3) ropivacaine with both dexamethasone and dexmedetomidine. Neither the children, parents, nor the clinical staff assessing pain will know which medication was given.

The goal of this study is to determine whether the combination of dexamethasone and dexmedetomidine provides longer pain relief and reduces the need for additional pain medication compared with either medication alone. The results may help identify the most effective and safest strategy for improving postoperative comfort in pediatric patients receiving regional anesthesia.

DETAILED DESCRIPTION:
Popliteal sciatic nerve block is frequently used in pediatric anesthesia to provide effective pain control for surgical procedures involving the lower leg, ankle, and foot. Although ropivacaine alone offers good analgesia, its duration is limited, and additional medications (adjuvants) are often added to prolong the effect of the block. Two commonly used adjuvants are dexamethasone, a corticosteroid, and dexmedetomidine, an alpha-2 adrenergic agonist. Each of these medications has been shown to extend the duration of analgesia, but it remains unclear whether combining them provides an additive or potentially synergistic benefit.

This randomized, double-blinded, controlled clinical trial will compare three perineural adjuvant strategies: dexamethasone, dexmedetomidine, and their combination. All participants will receive a single-shot popliteal sciatic nerve block with 0.2% ropivacaine. Children will then be randomized into one of three treatment arms:

1. ropivacaine with perineural dexamethasone,
2. ropivacaine with perineural dexmedetomidine, or
3. ropivacaine with a perineural combination of dexamethasone and dexmedetomidine. Pain scores, block duration, opioid use, and recovery parameters will be assessed by trained observers who are blinded to group assignment. The primary aim is to determine whether the combination of dexamethasone and dexmedetomidine leads to superior analgesia compared with either drug alone. Secondary aims include evaluating the time to first rescue analgesia, total postoperative opioid requirements, behavioral pain scores (e.g., FLACC), adverse events, and early functional recovery.

This study seeks to provide high-quality evidence to guide the optimal choice of perineural adjuvants in pediatric regional anesthesia and may help establish best-practice recommendations for improving postoperative comfort and safety in children undergoing lower-limb surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 12 years.
* Scheduled for elective unilateral lower limb surgery (foot, ankle, or distal lower leg) under general anesthesia with a popliteal sciatic nerve block planned for postoperative analgesia.
* ASA physical status I-III.
* Ability of parents or legal guardians to understand the study procedures and provide written informed consent.
* Child and parents/guardians available for telephone follow-up at 1 week and 1 month after surgery.

Exclusion Criteria:

* Refusal of the parents/legal guardians to provide informed consent or refusal of the child to cooperate with anesthesia or study procedures.
* Known allergy or hypersensitivity to ropivacaine, dexamethasone, dexmedetomidine, or any component of the study medications.
* Pre-existing neurological deficit or neuromuscular disease affecting the lower limbs (motor or sensory).
* Coagulopathy or current therapeutic anticoagulation that contraindicates regional anesthesia.
* Local infection, inflammation, or skin lesions at the planned block site.
* Severe cardiac, hepatic, renal, or respiratory disease that, in the investigator's opinion, increases the risk of study participation.
* History of clinically significant arrhythmias, severe bradycardia, or second/third degree atrioventricular block not treated with a pacemaker.
* Developmental delay or severe cognitive impairment that precludes reliable pain assessment or follow-up.
* Chronic use of opioid analgesics or sedatives (≥ 2 weeks of daily use before surgery).
* Participation in another interventional clinical trial within the last 30 days.
* Any other condition considered by the investigator to interfere with protocol adherence, safety monitoring, or reliable outcome assessment.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia | 0-24 hours postoperatively
  Time in hours from completion of the popliteal sciatic nerve block to the first administration of rescue analgesic medication. Rescue analgesia will be provided when the FLACC pain score is ≥ 4, or upon patient/parent request. This measure reflects the duration of effective postoperative analgesia provided by the nerve block.

SECONDARY OUTCOMES:
Total Opioid Consumption | 0-24 hours postoperatively
  Total amount of opioid rescue medication administered within the first 24 hours after surgery, converted to morphine milligram equivalents (MME). Includes all postoperative rescue doses documented in the anesthesia and nursing records.
FLACC Pain Scores at Rest | 2 hours postoperatively
  Pain intensity measured using the validated FLACC (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Assessments will be performed by trained, blinded observers.
FLACC Pain Scores at Rest | 4 hours postoperatively
  Pain intensity measured using the validated FLACC (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Assessments will be performed by trained, blinded observers.
FLACC Pain Scores at Rest | 8 hours postoperatively
  Pain intensity measured using the validated FLACC (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Assessments will be performed by trained, blinded observers.
FLACC Pain Scores at Rest | 12 hours postoperatively
  Pain intensity measured using the validated FLACC (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Assessments will be performed by trained, blinded observers.
FLACC Pain Scores at Rest | 24 hours postoperatively
  Pain intensity measured using the validated FLACC (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Assessments will be performed by trained, blinded observers.
FLACC Pain Scores During Movement | 2 hours postoperatively
  Pain scores assessed during standardized gentle movement of the operated limb using the FLACC scale (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Movement will be performed by a physiotherapist or trained nurse.
FLACC Pain Scores During Movement | 4 hours postoperatively
  Pain scores assessed during standardized gentle movement of the operated limb using the FLACC scale (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Movement will be performed by a physiotherapist or trained nurse.
FLACC Pain Scores During Movement | 8 hours postoperatively
  Pain scores assessed during standardized gentle movement of the operated limb using the FLACC scale (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Movement will be performed by a physiotherapist or trained nurse.
FLACC Pain Scores During Movement | 12 hours postoperatively
  Pain scores assessed during standardized gentle movement of the operated limb using the FLACC scale (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Movement will be performed by a physiotherapist or trained nurse.
FLACC Pain Scores During Movement | 24 hours postoperatively
  Pain scores assessed during standardized gentle movement of the operated limb using the FLACC scale (Face, Legs, Activity, Cry, Consolability) pain scale. Scores range from 0 (no pain) to 10 (severe pain). Movement will be performed by a physiotherapist or trained nurse.
Incidence of Adverse Events | 0-24 hours postoperatively
  Number of participants experiencing adverse events possibly related to the block or adjuvants, including excessive sedation, bradycardia, hypotension, local anesthetic systemic toxicity, injection-related complications, prolonged motor block, postoperative nausea or vomiting, or unexpected behavioral responses.
Incidence of Persistent Sensory or Motor Deficit (Nerve Injury Screening) | 1 week postoperatively
  Screening for signs of persistent sensory or motor dysfunction potentially related to the popliteal sciatic nerve block or perineural adjuvants. Follow-up will be conducted through structured telephone interviews with parents or guardians at 1 week and 1 month postoperatively. The assessment will include questions regarding persistent numbness, tingling, altered sensation, weakness of ankle or toe movement, gait abnormalities, or any parental concerns suggestive of nerve dysfunction. If abnormalities are reported, an in-person neurological examination will be offered. This measure assesses the potential impact of perineural dexamethasone, dexmedetomidine, or their combination on nerve integrity.
Incidence of Persistent Sensory or Motor Deficit (Nerve Injury Screening) | 1 month postoperatively
  Screening for signs of persistent sensory or motor dysfunction potentially related to the popliteal sciatic nerve block or perineural adjuvants. Follow-up will be conducted through structured telephone interviews with parents or guardians at 1 week and 1 month postoperatively. The assessment will include questions regarding persistent numbness, tingling, altered sensation, weakness of ankle or toe movement, gait abnormalities, or any parental concerns suggestive of nerve dysfunction. If abnormalities are reported, an in-person neurological examination will be offered. This measure assesses the potential impact of perineural dexamethasone, dexmedetomidine, or their combination on nerve integrity.

CONTACTS AND LOCATIONS:
Overall Officials: MAlgorzata Reysenr, MD PhD, Study Chair — Poznań University of Medicla Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
the primary and secondary outcomes will be made available to qualified researchers upon reasonable request. Shared data will include demographic information, details of the nerve block, intraoperative variables, postoperative pain scores, time to first rescue analgesia, opioid consumption, adverse events, and follow-up information regarding sensory or motor deficits. No direct identifiers or protected health information will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data and supporting documents will become available 12 months after publication of the primary results and will remain available for 5 years.
Access Criteria: Researchers must submit a methodologically sound proposal describing the planned use of the data. Requests will be reviewed by the study's principal investigators. Data will be shared only after signing a data access agreement and will be transferred using secure, password-protected methods.